CLINICAL TRIAL: NCT05139264
Title: GLADS Study: Glucose, Activity, Diet, & Sleep Assessment Study
Brief Title: Glucose, Activity, Diet, & Sleep Assessment Study
Acronym: GLADS
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Blandine Laferrere, Professor of Medicine, Columbia University
Other Study IDs: AAAT6779
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Metabolism Disorder, Glucose
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Observation of diet, physical activity, sleep and interstitial glucose

SUMMARY:
GLADS is a cross-sectional, observational study assessing free-living diet, physical activity, sleep, and glucose profile over a 2-week period in healthy adult men and women.

DETAILED DESCRIPTION:
Monitoring free-living lifestyle behaviors can provide important information on behavioral determinants of health. New technologies have improved accessibility of ambulatory assessment of diet, biomarkers, physical activity, and sleep. The study will assess the effects of free-living diet assessed by questionnaire and sleep and physical activity measured by actigraphy on interstitial glucose measured by continuous glucose monitoring in healthy adult men and women over a 2-week period.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 y old
* In possession of a smartphone
* English speaking
* Live in New York City metro area

Exclusion Criteria:

* Active food intake disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult men and women willing to record food intake with their smartphone, complete online questionnaires, and wear body sensors to measure physical activity, sleep, and glucose.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Glucose | 2 weeks
  Mean, fasting, post-prandial measured by continuous glucose monitoring

SECONDARY OUTCOMES:
Sleep duration | 2 weeks
  Measured by actigraphy
Sleep fragmentation | 2 weeks
  Measured by actigraphy
Diet composition | 2 weeks
  Carbohydrates, fats, proteins assessed by dietary recall

CONTACTS AND LOCATIONS:
Overall Officials: Blandine Laferrere, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Russ Berrie Medical Science Pavilion, New York, New York, United States